CLINICAL TRIAL: NCT03929471
Title: Target Weight Correction and Vascular Stiffness in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00086730
Record Dates: First submitted 2019-04-12; First posted 2019-04-26 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Fluid Overload; Vascular Stiffness
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients to be subjected to a fluid overload correction protocol.
  Interventions: Other: Target weight correction protocol
- Control group (No Intervention): Patient will be followed but no fluid overload correction protocol will be applied.

INTERVENTIONS:
Other: Target weight correction protocol — The intervention group will undergo target weight correction process based on time averaged fluid overload measurement (by bio-impedance).
  Arms: Intervention group

SUMMARY:
Title of the study: Target weight correction and vascular stiffness in hemodialysis patients Study design: Randomized clinical trial in the study centre at two locations

Applied medical device:

1. Body Composition Monitor' (BCM, Fresenius) to measure fluid volume overload.
2. Arteriograph 24 (Tensiomed, Budapest, Hungry) to assess vascular stiffness before, during and after the intervention.

Study hypothesis: A protocolized adjustment of target weight guided by bio-impedance spectroscopy will improve fluid status, systolic and diastolic blood pressure, and reduce the arterial wall stiffness without increasing the prevalence of intradialytic hypotension.

Aim of the study:

1. To demonstrate improvement in fluid status by a target weight correction protocol which applies BCM measurements.
2. To demonstrate that better fluid volume control is associated with a) improvement in vascular health as assessed by pulse wave velocity and augmentation index and b) reduction in antihypertensive medications use.
3. To show that this approach does not lead to more episodes with intradialytic hypotension.

The number of patients: 70 patients

DETAILED DESCRIPTION:
This study proposal is looking at the application of an accurate assessment of fluid status in hemodialysis (HD) patients to correct fluid overload. Patients undergoing hemodialysis suffer from the inability to maintain their normal body fluids and have a high probability to develop hypertension at initiation of dialysis (1). Long-standing fluid overload is no longer linked solely to high blood pressure, but also to vascular dysfunction and heart failure (1). Fluid overload is estimated based on the amount of fluids available outside the cells (extracellular fluid volume, ECFV). Thus, determination of the right amount of fluid removal during the dialysis depends on the weight of the patient when the ECFV is normal (referred to as Target Weight, TW). Essentially, TW is assessed by routine clinical judgment, for example, leg and hands swelling (edema), elevation in blood pressure and the expansion of the external jugular vein. Unfortunately, this clinical judgment is not reliable to assess fluid status (2, 3); hence, overestimation of TW occurs and leads to fluid overload. Current technology allows assessing fluid overload accurately by using bio-impedance, a non-invasive method that can be easily used in the HD setting. Despite this, very few studies have been reported where a systematic approach was followed to use bio-impedance to correct a TW that has been set too high, with the ultimate goal to correct fluid overload. Therefore, this study aims to provide better fluid control through an intervention to improve fluid status toward normovolemia by using bio-impedance assessment of fluid overload rather than clinical judgments. First, the fluid status will be measured in all study participants by multifrequency bio-impedance using a 'Body Composition Monitor' (BCM, Fresenius). Second, we will divide the study subjects into two groups; the control group which will initially receive standard conventional therapy (no intervention) for 3 months, and the intervention group will undergo by BCM measurements and integrated TW correction protocol for 3 months. Third, after three months, the control group will also involve in the same TW correction adjustment. The Primary outcome is improvement in fluid status towards normovolemia (<1.1 L fluid overload). Secondary outcomes are a) improvement in vascular health as assessed by pulse wave velocity and augmentation index and b) a decrease in the use of antihypertensive medications. Altogether, an optimized fluid status via implemented fluid management plan will provide better control of fluid overload, blood pressure, and improvement in vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) outpatients on 3-4 times per week HD sessions for at least 6 weeks with a life expectancy >6 months.
* Fluid overload ≥1.1L.
* Medically stable patient.
* Minimum of 3 hours of dialysis per session.

Exclusion Criteria:

* Pregnancy or lactation.
* Declined informed consent.

  * Patients with cognitive dysfunction.
  * Severe life-limiting Comorbidities (malignant tumour, tuberculosis,....)
  * Surgery within six weeks of the study.
  * Nocturnal dialysis patients.
  * Patients expected to receive a transplant or move to another center within the duration of the study.
  * Patients with arteriovenous fistula issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Fluid volume | through the study completion, an average of 6 months
  Improvement in fluid status towards normovolemia (<1.1 L fluid overload)

SECONDARY OUTCOMES:
Pulse wave velocity | Through the study completion, an average of 6 months
  Improvement in pulse wave velocity (millimetre/second)-one of vascular stiffness measurements
Augmentation index | Through the study completion, an average of 6 months
  Improvement in augmentation index (%)-one of vascular stiffness measurements
Anti hypertensive medications use | Through the study completion, an average of 6 months
  Reduction in the number of anti hypertensive medications use.

OTHER OUTCOMES:
Intradialytic hypotensive episodes (IDH) | Through the study completion, an average of 6 months
  The intervention will not lead to IDH episodes that happen during dialysis treatment. Such episodes including cramps, hypotension, and dizziness.

CONTACTS AND LOCATIONS:
Overall Officials: Branko Braam, MD PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No